CLINICAL TRIAL: NCT01259453
Title: Hepatitis B Vaccination Through Syringe Exchange Programs: A Randomized, Controlled Trial of Vaccination Schedules
Acronym: HVS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: DePaul University (Other); Hispanic Health Council, Inc. (Other); Case Western Reserve University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Robert Heimer, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0005011791; 5R01DA014502 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis B vaccination; Syringe exchange programs; Injection drug users; Hepatitis B prevention through vaccination
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard vaccination schedule (Active Comparator): Standard dosing at 0, 1, and 6 months
  Interventions: Biological: Vaccination to prevent hepatitis B virus infection
- Accelerated Schedule (Active Comparator): Accelerated dosing at 0, 1, and 2 months
  Interventions: Biological: Vaccination to prevent hepatitis B virus infection

INTERVENTIONS:
Biological: Vaccination to prevent hepatitis B virus infection — Standard dosing with Twinrix; comparison of standard and acceleration dosing schedule

SUMMARY:
The investigators seek to provide immunization for individuals who are at high risk of contracting hepatitis B virus (HBV) infection because of their illicit drug use. The investigators will be using the syringe exchange programs (SEPs) in Hartford and Bridgeport, CT and Chicago, IL to contact high risk individuals and refer them for vaccination. The primary purpose of the study is to compare the standard schedule of hepatitis B vaccination at 0, 1, and 6 months to an accelerated schedule of vaccination at 0, 1, and 2 months. The investigators hypothesize that the accelerated scheduling will result in improved completion rates without significant loss in vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate evidence of recent injection drug use (injection stigmata),
* 18 years of age or older,
* Screened for and found susceptible to HBV
* Able to provide informed consent.

Exclusion Criteria:

* Evidence of intoxication that prevented provision of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2003-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Vaccine Efficacy | 8 months from study enrollment

SECONDARY OUTCOMES:
Vaccine completion rate | 8 months from study enrollment
Association of exchange status with completion | 8 months from study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Heimer, Ph.D., Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Hispanic Health Council, Hartford, Connecticut
  - DePaul University, Chicago, Illinois
  - Case Western Reserve Universtiy, Cleveland, Ohio

REFERENCES:
- [Result] Hu Y, Grau LE, Scott G, Seal KH, Marshall PA, Singer M, Heimer R. Economic evaluation of delivering hepatitis B vaccine to injection drug users. Am J Prev Med. 2008 Jul;35(1):25-32. doi: 10.1016/j.amepre.2008.03.028. PMID 18541174